CLINICAL TRIAL: NCT00736606
Title: A Phase I, Single Centre, Open-Label Study to Assess the Pharmacokinetics of Both AZD9056 (Steady State) and Simvastatin (Single Dose) When Co-Administered in Healthy Volunteers
Brief Title: A Study to Assess Co-Administered AZD9056 (Steady State) and Simvastatin (Single Dose) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton, MD, PhD, Medical Science Director, AstraZeneca R&D Alderely Park
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1520C00008; EudraCt nr 2008-003626-41
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Volunteers
Keywords: simvastatin; AZD5672
MeSH Terms: interventions — Simvastatin; AZD9056

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Experimental): simvastatin
  Interventions: Drug: simvastatin
- Period 2 (Experimental): simvastatin + AZD9056
  Interventions: Drug: AZD9056 + simvastatin

INTERVENTIONS:
Drug: simvastatin — One single dose of 40mg
  Other Names: Zocor
  Arms: Period 1
Drug: AZD9056 + simvastatin — AZD9056: 400 mg od, 8 days simvastatin: one single dose of 40 mg on day 7
  Other Names: Zocor
  Arms: Period 2

SUMMARY:
The purpose of the study is to assess the pharmacokinetics of both AZD9056 (steady state) and simvastatin (single dose) when co-administered in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Male or female healthy subjects. Females should not be of childbearing potential
* Clinically normal physical and laboratory findings as judged by the investigator, including negative test results for drug-of-abuse, alcohol and cotinine at the Screening Visit and/or admission (Day -1) of each study period, and negative test results

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subject's ability to participate
* Known allergy to simvastatin (or other statins) or previous complications to simvastatin therapy.
* Participation in a clinical study involving an investigational product within 5 half-lives of active moieties of the last dose of investigational product or 3 months prior to first dosing (whichever is longer).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during study periods

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Rod Hepburn, Study Director — AstraZeneca R&D, Charnwood, UK; Maura Fallon, Principal Investigator — PAREXEL Clinical Pharmacology Research Unit
Locations (1):
- Research Site, Berlin, Germany